CLINICAL TRIAL: NCT01971762
Title: Staphylococcus Aureus Bacteremia: Impact of an Intervention Program in Improving the Clinical Management and Review of the Clinical and Molecular Epidemiology
Status: Completed | Type: Observational
Sponsor: Fundación Pública Andaluza Progreso y Salud (Other)
Responsible Party: Sponsor
Organization: Andalusian Network for Design and Translation of Advanced Therapies (Other)
Other Study IDs: FPS-STA-2011-01
Record Dates: First submitted 2013-10-18; First posted 2013-10-29 (Estimated); Last update posted 2014-12-05 (Estimated); Status verified 2013-11

CONDITIONS: Staphylococcus Aureus Bacteremia
Keywords: multiresistant bacteremia; bacteremia management; blood culture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients diagnosed bacteremia by S. aureus
  Interventions: Behavioral: Follow recommendations based on scientific evidence to S. aureus bacteremia management; Behavioral: Not to follow recommendations based on scientific evidence to S. aureus bacteremia management

INTERVENTIONS:
Behavioral: Follow recommendations based on scientific evidence to S. aureus bacteremia management
Behavioral: Not to follow recommendations based on scientific evidence to S. aureus bacteremia management

SUMMARY:
Staphylococcus aureus bacteremia: impact of an intervention program in improving the clinical management and review of the clinical and molecular epidemiology.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 14
* Clinical significant bacteremia by S. aureus
* Patient hospitalized

Exclusion Criteria:

* Non clinical significant bacteremia
* Ambulatory patient
* End-of-life patients

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients diagnosed bacteremia by S. aureus attended in participating centers will be included
Sampling Method: Non-Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2011-04; Primary Completion 2011-10 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
The overall target is to assess if the implementation of an active intervention program improves clinical management of the disease, according to existing recommendations. | 6 months
  Identify evidence-based quality-of-care indicators (QCIs) for the management of Staphylococcus aureus bacteremia (SAB).
  See secondary objective for the definitions of QCIs

SECONDARY OUTCOMES:
Follow-up blood cultures performance of control blood culture 48-96h. | 6 months
  Description:Performance of control blood cultures 48-96 h after antimicrobial therapy was started regardless of clinical evolution
  Formula:Patients with follow-up blood culture collected×100/Patients alive at 96h.
Early source control | 6 months
  Description: Removal of nonpermanent vascular catheter whenever the catheter was suspected or confirmed as the source of SAB, or drainage of an abscess in <72 h.
  Formula: Patients in which the amenable source was removed in<72h×100/Patients with source amenable of removal/drainage
Echocardiography in patients with clinical indications | 6 months
  Description: Performance of echocardiography in patients with complicated bacteremia or predisposing conditions for endocarditis.
  Formula: Patients with echocardiography×100/Patients with complicated bacteremia or predisposing condition for endocarditis,alive at 96h
Early use of IV cloxacillin for meticillin susceptible Staphylococcus aureus as definitive therapy | 6 months
  Description: Definitive therapy with intravenous cloxacillin (at least 2 g every 6 h or adjusted based on renal function in renal failure) in cases of methicillin-susceptible strains (allergic patients excluded). Treatment should be started within the first 24 h after methicillin sensitivity was available. For hemodialysis patients, cefazolin 2 g after each hemodialysis session was acceptable
  Formula: Definitive therapy with IV cloxacillin×100/nonallergic Patients with methicillin-susceptible isolates.
Adjustment of vancomycin dose according to trough levels. | 6 months
  Description: Measurement of trough levels of vancomycin in patients treated for at least 3 d with this antibiotic and adjustment of dose in order to achieve plasma trough levels between 15 and 20 mg/L in survivors
  Formula: Patients with trough level of vancomycin determined and dose adjusted×100/Patients treated with vancomycin,at 3d.
Treatment duration according to the complexity of infection. | 6 Months
  Description: Duration of antimicrobial therapy of at least 14 d for uncomplicated bacteremia and 28 d for complicated bacteremia. Sequential oral treatment with fluoroquinolone plus rifampin, trimethoprim-sulfamethoxazole, or linezolid was considered accepted in selected case.
  Formula:Patients with appropriate duration of therapy×100/P alive at 14 or 28d in uncomplicated or complicated bacteremia

CONTACTS AND LOCATIONS:
Overall Officials: Jesús Rodríguez-Baño, Principal Investigator — Hospital Universitario Virgen Macarena
Locations (16):
- Spain (16):
  - Hospital de Puerto Real, Puerto Real, Cádiz
  - Hospital Costa del Sol, Marbella, Málaga
  - Hospital de Torrecárdenas, Almería
  - Hospital de barcelona - SCIAS, Barcelona
  - Hospital de Cruces, Bilbao
  - Hospital Puerta del Mar, Cadiz
  - Hospital Reina Sofía, Córdoba
  - Hospital Virgen de las Nieves, Granada
  - Hospital Juan Ramón Jiménez, Huelva
  - Hospital de San Pedro, Logroño
  - Hospital Carlos Haya, Málaga
  - Hospital Virgen de la Victoria, Málaga
  - Hospital de la Arrixaca, Murcia
  - Hospital de Valdecillas, Santander
  - Hospital Universitario Virgen de la Macarena, Seville
  - Hospital Virgen de Valme, Seville

REFERENCES:
- [Result] Lopez-Cortes LE, Del Toro MD, Galvez-Acebal J, Bereciartua-Bastarrica E, Farinas MC, Sanz-Franco M, Natera C, Corzo JE, Lomas JM, Pasquau J, Del Arco A, Martinez MP, Romero A, Muniain MA, de Cueto M, Pascual A, Rodriguez-Bano J; REIPI/SAB group. Impact of an evidence-based bundle intervention in the quality-of-care management and outcome of Staphylococcus aureus bacteremia. Clin Infect Dis. 2013 Nov;57(9):1225-33. doi: 10.1093/cid/cit499. Epub 2013 Aug 8. PMID 23929889